CLINICAL TRIAL: NCT03307070
Title: Adapted Cognitive Behavioral Treatment for Depression in Patients With Moderate to Severe Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Lauren Fisher, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002823
Record Dates: First submitted 2017-10-04; First posted 2017-10-11 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Depressive Disorder, Major; Brain Injuries, Traumatic | interventions — Cognitive Behavioral Therapy; Whole-Body Irradiation

STUDY DESIGN:
Intervention Model Description: The study is a randomized, waitlist controlled trial. All participants randomized to waitlist were offered the opportunity to receive the intervention after completion of the waitlist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Active Comparator): Participants who are randomized to begin the Cognitive Behavioral Therapy for individuals with TBI immediately after screening. This treatment is a version of Cognitive Behavioral Therapy (CBT) adapted specifically for patients who have experienced a moderate to severe Traumatic Brain Injury (TBI).
  Interventions: Behavioral: Cognitive Behavioral Therapy for individuals with TBI
- Waitlist Control (Other): Participants who are randomized to be put on a waitlist after screening. After 12 weeks of being on the waitlist, participants will be offered the Cognitive Behavioral Therapy for individuals with TBI
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for individuals with TBI — Cognitive Behavioral Therapy for depression that has been adapted for a population who has experienced a moderate to severe Traumatic Brain Injury. This is a 12 week long treatment for depression with weekly visits that challenges negative thoughts and behaviors. This version has been specifically developed for the study to account for specific cognitive needs of individuals who have experienced a moderate to severe TBI.
  Arms: Active Group
Other: Waitlist Control — Participants will be randomized to a waitlist. They will attend biweekly study sessions for 12 weeks to track progress, but will receive their treatment as usual.
  Arms: Waitlist Control

SUMMARY:
Cognitive behavioral therapy for major depressive disorder (MDD) was adapted for individuals with moderate to severe traumatic brain injury (TBI) (CBT-TBI). A structured, treatment manual was developed.

The primary aim is to evaluate the acceptability and tolerability of, and adherence to, CBT-TBI in a randomized waitlist-controlled, 12-week pilot trial (N=40).

The exploratory aim is to evaluate the potential efficacy of CBT-TBI for MDD in the randomized pilot trial (N=40) and possible moderators and mediators of outcome.

DETAILED DESCRIPTION:
The primary aim of this study is to develop a highly acceptable, manualized treatment (CBT-TBI) for MDD in patients with moderate to severe TBI. Initial feasibility data from a small, open pilot will inform the randomized controlled trial. Primary analyses will examine feasibility and acceptability of the intervention. The investigators will then pilot test the efficacy of the intervention to reduce depressive symptoms (IDS-C) after 12 weeks compared to a waitlist control group.

The proposed study involves the following points of contact: (1) Obtaining informed consent and screening (may be broken up into multiple visits), (2) biweekly clinician assessments of depressive and neuropsychiatric symptoms (weeks 2, 4, 6, 8, 10), (3) weekly self-report assessments of depressive symptoms for those receiving the intervention, (4) 12 weekly individual CBT-TBI sessions for those randomized to the intervention, (5) a comprehensive assessment at week 12 (primary endpoint), which includes the neuropsychological battery, and (6) a 3-month follow-up assessment for those who received the intervention. The week 12 visit can be split into two parts, with the neuropsychological assessment occurring during the second part, in order to accommodate subjects' potential limitations due to fatigue. Procedures for this study were all conducted remotely after March 17, 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 and older
2. English language proficiency
3. Ability to provide written, informed consent; OR consent provided by legally authorized representative with assent from subject
4. Ability to see and hear (hearing or visual loss cannot impair ADLs or in-room conversation)
5. Has access to a smartphone/tablet/computer with internet and video capabilities for virtual sessions
6. Having been hospitalized for moderate to severe TBI that occurred at least 3 months prior to study entry
7. Meeting ANY ONE of the following severity criteria, as documented in electronic medical record (EPIC) or available outside records:

   1. GCS 3-12 with GCS motor score ≤ 5 within 4 hours after injury
   2. GCS 3-12 with GCS motor score =6 within 4 hours after injury AND documented intracranial abnormalities on imaging
   3. GCS 13-15 within 4 hours after injury AND documented intracranial abnormalities on imaging
   4. Loss of consciousness (LOC) > 30 min.
   5. Post-traumatic amnesia (PTA) > 24 hours
8. Out of PTA at the time of enrollment (GOAT>75)
9. Clinically significant depressive symptoms: meets criteria for Major Depressive Episode on the MINI or has a total score ≥ 23 on the Inventory of Depressive Symptomatology - Clinician rated (IDS-C)

Exclusion Criteria:

1. Uncontrolled medical illness
2. Behavioral dyscontrol, defined as the presence of verbally or physically aggressive behavior in the past month, as evidenced in medical records, pre-screening interviews, or observed by any study staff
3. Presents with PTSD as the primary diagnosis, as determined by a clinician
4. Substance use disorder, moderate or severe, within the past 6 months
5. Has bipolar disorder, a primary psychotic disorder or current psychotic symptoms, or acute suicidality or homicidality
6. Currently receiving regular (≥ 2 times/ mo.) psychosocial treatment for depression
7. Has participated in CBT for depression within the past 6 months
8. Individuals with history of dementia or severe cognitive impairment that is not related to TBI (e.g., cognitive impairment requiring assistance with basic activities of daily living, such as getting ready in the morning)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-23 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Feasibility - retention/completion rates | 12 weeks
  For examining the feasibility of treatment with CBT-TBI, descriptive analyses will be conducted to assess participants' retention/completion rates across study visits.
Feasibility - drop out rates | 12 weeks
  For examining the feasibility of treatment with CBT-TBI, descriptive analyses will be conducted to assess participants' drop-out rates across study visits.
Feasibility - randomization, recruitment rates | 12 weeks
  For examining the feasibility of treatment with CBT-TBI, descriptive analyses will be conducted to assess rate of recruitment and randomization (number randomized/number consented).
Acceptability - satisfaction with treatment | 12 weeks
  Descriptive analyses will be conducted to assess participants' satisfaction with CBT-TBI (Satisfaction with Therapy and Therapist Scale - Revised).

SECONDARY OUTCOMES:
Efficacy - Treatment Response [Inventory of Depressive Symptomatology - Clinician Rated (IDS-C)] (Exploratory Aim) | 12 weeks
  The IDS-C is a 30-item clinician rated scale that assesses severity of depression. Scores range from 0 to 84, with higher scores indicative of greater depression severity.
  Descriptive analyses will be performed for percentage of responders (defined as 50% improvement on the IDS-C total) and remitters (≤6 on IDS-C total) at the end of treatment. The percent of responders and remitters in each group will be computed in order to estimate an effect size for a larger trial.
Efficacy - Treatment Response [Inventory of Depressive Symptomatology - Clinician Rated (IDS-C)] (Exploratory Aim) | 12 weeks
  The IDS-C is a 30-item clinician rated scale that assesses severity of depression. Scores range from 0 to 84, with higher scores indicative of greater depression severity.
  Change in depressive severity (IDS-C total) scores from baseline to post-treatment will also be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Fisher, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fisher LB, Tuchman S, Curreri AJ, Markgraf M, Nyer MB, Cassano P, Iverson GL, Fava M, Zafonte RD, Pedrelli P. Transitioning From In-Person to Remote Clinical Research on Depression and Traumatic Brain Injury During the COVID-19 Pandemic: Study Modifications and Preliminary Feasibility From a Randomized Controlled Pilot Study. JMIR Form Res. 2021 Dec 1;5(12):e28734. doi: 10.2196/28734. PMID 34662285

DOCUMENTS (2):
  • Study Protocol (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT03307070/Prot_004.pdf
  • Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT03307070/SAP_005.pdf